CLINICAL TRIAL: NCT02911961
Title: Serum Acetaminophen-Cysteine (APAP-CYS) Adduct Concentrations in Subjects Expected to Develop Aminotransferase Elevations With Liver-Directed Therapy Intended to Treat Hepatic Tumors
Brief Title: APAP-CYS Protein Adduct Concentrations in Patients With Liver-Directed Therapy Intended to Treat Hepatic Tumors
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to lack of enrollment and organizational desire to focus recruitment efforts on other studies.
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry); University of Colorado, Denver (Other); Rocky Mountain Poison and Drug Center (Unknown)
Responsible Party: Principal Investigator, Kennon Heard, Principal Investigator, Denver Health and Hospital Authority
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 16-0031
Record Dates: First submitted 2016-08-17; First posted 2016-09-23 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Acetaminophen Exposure
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acetaminophen (Experimental): Subjects will take extra strength acetaminophen (4g/day) for the three days prior to the embolization procedure.
  Interventions: Drug: Acetaminophen
- Observational - No Acetaminophen (No Intervention): Subjects will take no acetaminophen containing products prior to the embolization procedure.

INTERVENTIONS:
Drug: Acetaminophen — 1 gram acetaminophen 4 times a day with at least 6 hour intervals between doses for the 3 days prior to the embolization procedure.
  Other Names: Tylenol
  Arms: Acetaminophen

SUMMARY:
The objective of this study is to provide preliminary data to describe serum acetaminophen-cysteine protein adduct (APAP-CYS) concentrations following therapeutic doses of acetaminophen in the setting of non-acetaminophen induced liver injury. This study will utilize hepatic embolization as a model of hepatic injury.

DETAILED DESCRIPTION:
Acetaminophen-cysteine protein adducts (APAP-CYS) are formed when acetaminophen is oxidized by CYP 2E-1. When hepatocytes die, these proteins are released into the serum and can be detected. APAP-CYS can therefore be an experimental biomarker of acetaminophen exposure. It is possible that massive necrosis of hepatocytes that contain APAP-CYS from therapeutic doses of acetaminophen can be misinterpreted as acetaminophen overdose as the cause of liver injury. This study aims to describe serum APAP-CYS concentrations in patients taking a therapeutic dose of acetaminophen who develop a liver injury from a cause other than acetaminophen. This study will seek to enroll subjects undergoing a hepatic embolization procedure to treat a secondary liver tumor. This procedure is a reproducible model of non-acetaminophen induced hepatic injury. A small number of subjects who are otherwise eligible to participate but are unwilling to take acetaminophen will be offered participation in the observational arm of the study. They will undergo the same assessments with the exception of acetaminophen dosing. Subjects willing to take acetaminophen will be asked to take extra strength acetaminophen (4g/day) for the 3 days prior to their embolization procedure. All subjects will be asked to keep a detailed medication diary for the three days prior and up to their embolization procedure. Blood samples for the measurement of APAP-CYS concentrations and markers of liver function will be collected prior to acetaminophen dosing, prior to the embolization procedure, and at several time points after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any gender or ethnic background who are between 21 and 80 years old
* Subjects who are able to provide written, informed consent
* Subjects with secondary liver cancer
* Subjects undergoing portal vein or bland embolization for the treatment of secondary hepatic tumor
* Subjects who are willing to have their blood drawn at least 12 times for study purposes
* Subjects who agree to stay for ~18-21 hours after being discharged from the Department of Radiology for research purposes
* Subjects who agree to refrain from using acetaminophen, other than the study drug, during the dosing phase through a minimum of 5 days post-procedure
* Subjects who agree to consume less than 3 alcoholic drinks per day while taking study drug (acetaminophen group only)
* Subjects who are willing to complete a study diary for 3 days prior to and the day of the procedure
* Subjects who will be in the Denver metro area for the duration of the study

Exclusion Criteria:

* Subjects with known cirrhosis
* Subjects with a history of moderate to severe anemia at screening as defined by:

  1. Moderate: Hemoglobin 8-9.5 g/dL
  2. Severe: Hemoglobin <8 g/dL
* Subjects with an ALT or AST greater than 200 IU/L at screening
* Subjects with a total bilirubin greater than 1.5 mg/dL at screening
* Subjects with an INR greater than 1.3 at screening
* Subjects with a platelet count less than 125 10^9/L at screening
* Subjects who are currently taking warfarin (acetaminophen group only)
* Subjects with anorexia nervosa (self-reported; acetaminophen group only)
* Subjects who weigh ≤50 kg at screening (acetaminophen group only)
* Subjects who adhere to a fasting type diet (self-reported; acetaminophen group only)
* Subjects with a known hypersensitivity or allergy to acetaminophen (acetaminophen group only)
* Subjects who are currently taking isoniazid (acetaminophen group only)
* Subjects who are currently taking disulfiram (acetaminophen group only)
* Subjects who are pregnant or breastfeeding (female participants only)
* Subjects who are currently enrolled in a clinical trial, have participated in a clinical trial within the 30 days prior to the procedure, or who plan to participate in a clinical trial during the 5 day post-procedure follow-up period

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
APAP-CYS Concentrations Over Time - Acetaminophen Group | 14 days
  To describe the course of APAP-CYS concentrations following hepatic embolization in subjects who receive 4 grams/day of acetaminophen for three days prior to the procedure

SECONDARY OUTCOMES:
APAP-CYS Concentrations Over Time - Non-Acetaminophen Group | 2 years
  To determine if subjects who report no exposure to acetaminophen prior to the procedure have detectable APAP-CYS concentrations
Relationship between APAP-CYS and other biochemical markers of liver function | 2 years
  To evaluate the relationship between APAP-CYS concentrations with aspartate aminotransferase (AST), alanine aminotransferase (ALT), and miRNA activity

CONTACTS AND LOCATIONS:
Overall Officials: Kennon Heard, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No